CLINICAL TRIAL: NCT02185521
Title: Hemodynamic Instability Rules Based Advisor: The Impact to Care With a New Predictive Indicator (HIRBA 2.0)
Brief Title: Hemodynamic Instability Index: The Impact to Care With a New Predictive Indicator
Acronym: HII
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initial main phase completed but recruitment rate was too slow to continue.
Sponsor: Philips Healthcare (Industry)
Collaborators: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2917-05-12-433
Record Dates: First submitted 2014-06-24; First posted 2014-07-09 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Shock; Hemodynamic Instability
Keywords: Hemodynamics; Medical Informatics
MeSH Terms: conditions — Shock | interventions — Patient Outcome Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- visible HII - patient assessment (Experimental): Clinical team from study unit will observe the Hemodynamic Instability Index created by the HIRBA 2.0 system for individual subjects randomized into HII group arm.
  If the HII value will cross the threshold, indicative of hemodynamic deterioration, subject from the study arm will receive intervention: clinical assessment.
  Interventions: Other: patient assessment

INTERVENTIONS:
Other: patient assessment — Patient clinician status assessment based on Hemodynamic Instability Indicator (HII) trend. The HII indicator combines existing data such as physiologic parameters (Heart Rate, HR; Blood Pressure, BP), laboratory measurements (Albumin; Hematocrit, HCT; Bicarbonate; White Blood Cell, WBC; Blood Urea Nitrogen, BUN), and ADT information (age). HII will be displayed on charting workstation (Workstation on Wheels, WOW). Nurse's role will be to observe the value of HII while accessing WOW desktop (during regular charting), interpret HII value, and share this information to the physician when indicative of potential patient hemodynamic instability to trigger patient clinical status assessment. This intervention is associated with Experimental Study Arm: visible HII.

SUMMARY:
Philips has developed a new algorithm, called Hemodynamic Instability Rules Based Advisor (HIRBA 2.0) system, for the prediction of hemodynamic instability in critically ill patients, who were not previously known to be at risk. This algorithm provides with the numerical index - Hemodynamic Instability Index (HII) and its trend which are calculated from existing real time data derived from patient's current hospital stay such as heart rate and blood pressure, labs, and Admission - Discharge- Transfer (ADT) data to help healthcare providers obtain information about patient's status and make clinical decisions.

The aim of the study is to determine if the patient clinical information, displayed in the form of HII, can prompt possible patient hemodynamic status change and trigger earlier clinical care team response. We hypothesize that this real-time information on hemodynamic instability and earlier clinical decision making will lead to reduced length of stay (LOS) and ICU mortality relative to standard care practice. Study will also identify if the use of the Philips new algorithm called Hemodynamic Instability Rules Based Advisor (HIRBA 2.0) can improve outcomes for patients admitted to the intensive care units (ICUs).

During this study, upon patient admission to the ICU clinical data collection will begin. Data that will be pulled during the study includes: vital signs, medications, reason for admission to the ICU, treatments that patient may receive.

Research subjects will not be asked to do anything as far as specific activities expected to be accomplished during study participation. Subjects will be involved in the study only during their stay in ICU. HII information will be visible to clinicians, taking care of this patient only during his/ her stay in the study unit.

Study team will collect patient information and have the ability to view the HII for subjects.

Once patient leaves the ICU the study team will collect information on the remainder of patient's hospital course including date of hospital discharge. All collected data will be then fully de-identified and released to Philips for analysis.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the study unit will be invited to participate in the study.
* Study subject has to stay in study unit for at least 12 hours.

Exclusion Criteria:

* Patients who were discharged from study unit earlier then 12 hours after admission.
* Patients who are or become dependent on extracorporeal membrane oxygenation (ECMO) support.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2016-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant V Bochicchio, MD, Principal Investigator — Washington University School of Medicine; Mitchell M Levy, MD, Principal Investigator — Alpert Medical School of Brown University, Rhode Island Hospital, Providence RI
Locations (2):
- United States (2):
  - Washington University in St. Louis School of Medicine, Department of Surgery, Section of Acute and Critical Care Surgery, St Louis, Missouri
  - Alpert Medical School of Brown University, Rhode Island Hospital, Medical Intensive Care Unit, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients admitted to the surgical, trauma and burn ICU were evaluated for inclusion/exclusion criteria. Those who met eligibility were approached for informed consent. Legally Authorized Representatives (LAR's) were approached for patients who were too injured or ill to participate in the informed consent process.
Pre-assignment Details: If a Legally Authorized Representative (LAR) consented on behalf of the participant and later the participant had the capacity to self-consent and decided not to participate in the study, the participant was dropped from the study.
Groups:
- Visible HII - Patient Assessment: Clinical team from study unit will observe the Hemodynamic Instability Index created by the HIRBA 2.0 system.
  If the HII value will cross the threshold, indicative of hemodynamic deterioration, subject from the study arm will receive intervention: clinical assessment.
  Patient assessment: Patient clinician status assessment based on HII trend. The HII indicator combines existing data such as physiologic parameters (HR, BP), laboratory measurements (Albumin, HCT, Bicarbonate, WBC, BUN), and ADT information (age). HII will be displayed on charting workstation (WOW). Nurse's role will be to observe the value of HII while accessing WOW desktop (during regular charting), interpret HII value, and share this information to the physician when indicative of potential patient hemodynamic instability to trigger patient clinical status assessment. This intervention is associated with Experimental Study Arm: visible HII.
Period: Overall Study
Arm/Group | Visible HII - Patient Assessment
Started | 127
Completed | 125
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Visible HII - Patient Assessment
Number analyzed (Participants) | 125
Age, Continuous [Mean (Full Range); unit: Years] | 56 [18 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 80
Treatment [Number; unit: participants]
  Intraveneous (IV) med (inotropes/pressors) | 57
  Intraveneous (IV) med weak | 16
  Fluid resuscitation | 97
  Packed Red Blood Cells (PRBC) | 69
  Any hemodynamic intervention | 83
  No hemodynamic interventions | 16
Surgical Type [Count of Participants; unit: Participants]
  Elective | 9
  Urgent/Emergent | 81
  N/A | 34
  Unknown | 1
Monitoring - Arterial line [Count of Participants; unit: Participants] | 92

OUTCOME MEASURES:

1. Primary Outcome: Intensive Care Unit (ICU) Length of Stay
Time Frame: From time of the study subject admission to the unit until the day of discharge of that same study subject from the unit, assessed up to 12 months.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Visible HII - Patient Assessment: Clinical team from study unit will observe the Hemodynamic Instability Index created by the HIRBA 2.0 system for individual subjects randomized into HII group arm.
  If the HII value will cross the threshold, indicative of hemodynamic deterioration, subject from the study arm will receive intervention: clinical assessment.
  patient assessment: Patient clinician status assessment based on HII trend. The HII indicator combines existing data such as physiologic parameters (HR, BP), laboratory measurements (Albumin, HCT, Bicarbonate, WBC, BUN), and ADT information (age). HII will be displayed on charting workstation (WOW). Nurse's role will be to observe the value of HII while accessing WOW desktop (during regular charting), interpret HII value, and share this information to the physician when indicative of potential patient hemodynamic instability to trigger patient clinical status assessment. This intervention is associated with Experimental Study Arm: visible HII.
Arm/Group | Visible HII - Patient Assessment
Number analyzed (Participants) | 125
days | 6.68 (9.57)

2. Secondary Outcome: Intensive Care Unit (ICU) Mortality
Time Frame: From date of randomization of the study subject until the date of ICU discharge, an average of 6.7 days..
Measure: Count of Participants; unit: Participants
Arm/Group | Visible HII - Patient Assessment
Number analyzed (Participants) | 125
Participants | 12

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Visible HII - Patient Assessment
All-Cause Mortality (participants affected / at risk) | 12/127
Serious Adverse Events (participants affected / at risk) | 0/127
Other Adverse Events (participants affected / at risk) | 0/127

LIMITATIONS AND CAVEATS:
Slow recruitment led to early termination of the study; generalizability to other ICU settings; lack of further analyses due to small sample size and data collected (timing of intervention, morbidity, cost reduction).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No